CLINICAL TRIAL: NCT05505864
Title: A Combined Health Action Process Approach and mHealth Intervention to Assess Sedentary Behaviour in Adults With Type 2 Diabetes - A Randomized Controlled Trial
Brief Title: Assessing Sedentary Behaviour in Adults With Type 2 Diabetes - A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University (Other)
Responsible Party: Principal Investigator, Siobhan Smith, Dr Harry Prapavessis, Principal Investigator, Western University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 120585
Record Dates: First submitted 2022-07-27; First posted 2022-08-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Sedentary Behavior; Diabetes Mellitus, Type 2; Adult ALL
MeSH Terms: conditions — Sedentary Behavior; Diabetes Mellitus, Type 2; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): * Participants in the intervention group will be asked to wear an ACTIVPAL4 at week 0, 5, and 11.
  * Participants in the intervention group will be asked to fill out questionnaires assessing key variable (demographics, sedentary behaviour, and quality of life) on the SEMA3 app at week 0, 2, 4, 6, and 12.
  * Participants in the intervention group will receive a one-on-one behavioural counselling session online through zoom at week 0 to create personalized action plans and coping strategies to reduce and break up sedentary behaviour. The participant will update these action plans and coping strategies at the end of week 2 and 4 on the SEMA3 app.
  * Participants in the intervention group will receive tailored text messages the day after receiving their one-on-one counselling session for a 6-week period.
  * Participants in the intervention will receive one-on-one qualitative interview on zoom at week 6 to explore participants overall experience engaging in the intervention.
  Interventions: Behavioral: Health Action Process Approach (HAPA)
- Control Group (No Intervention): * Participants in the control group will be asked to wear an ACTIVPAL4 at week 0, 5, and 11.
  * Participants in the control group will be asked to fill out questionnaires assessing key variable (demographics, sedentary behaviour, and quality of life) on the SEMA3 mobile app at week 0, 2, 4, 6, and 12.

INTERVENTIONS:
Behavioral: Health Action Process Approach (HAPA) — Health Action Process Approach (HAPA) using action planning and coping strategies to create health behaviour change
  Arms: Intervention Group

SUMMARY:
The purpose of this health behaviour change research study is to assist adults with T2D in achieving the Canadian 24-hour sedentary behaviour movement guidelines.

DETAILED DESCRIPTION:
Adults with type 2 diabetes (T2D) are less active and accumulate more sedentary behaviour (SB) than those without. Among adults with T2D, increased SB is associated with increased mortality after adjusting for physical activity. Canadian 24-hour SB movement guidelines recommend limiting SB to ≤8 hours, no more than 3 hours of recreational screen time, and breaking up long periods of SB as often as possible. Therefore, the purpose of this research study is for adults with T2D to achieve these SB Canadian 24-hour SB movement guidelines. To address this purpose, we will be conducting a six-week two-arm repeated measures randomized control trial. The intervention group will receive a theory-based behaviour change counselling session through zoom at week 0, mobile phone application at weeks 2 and 4 that encourage participants to create their own personal and specific action plans and coping strategies, and daily text messages that motivate participants to reduce and break up their SB. The control group will receive no intervention. The primary objective of the study is to reduce SB, while the secondary objectives are to break up SB, reduce screen time, improve quality of life, determine the perceptions towards the intervention, and validate the SB questionnaires. SB will be collected in the form of total daily SB, frequency of SB breaks, and duration of SB breaks. These variables will be measured through a SB and quality of life questionnaires that will be delivered through a downloadable mobile phone application. Outcome measures will be compared within and between groups to detect differences.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* diagnosed with type 2 diabetes
* access to a smart phone with internet connection
* be able to read, write, and speak in english

Exclusion Criteria:

* any medical or physical limitation that would prevent standing, stretching, and/or light physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Self-reported total sedentary behaviour | Measured at week 0.
  Measured by the modified sedentary behaviour questionnaire (SBQ). Where total daily sedentary behaviour ranges from 0 to 24 hours. Higher number of hours is worse.
Self-reported total sedentary behaviour | Measured at week 2.
  Measured by the modified sedentary behaviour questionnaire (SBQ). Where total daily sedentary behaviour ranges from 0 to 24 hours. Higher number of hours is worse.
Self-reported total sedentary behaviour | Measured at week 4.
  Measured by the modified sedentary behaviour questionnaire (SBQ). Where total daily sedentary behaviour ranges from 0 to 24 hours. Higher number of hours is worse.
Self-reported total sedentary behaviour | Measured at week 6.
  Measured by the modified sedentary behaviour questionnaire (SBQ). Where total daily sedentary behaviour ranges from 0 to 24 hours. Higher number of hours is worse.
Self-reported total sedentary behaviour | Measured at week 12.
  Measured by the modified sedentary behaviour questionnaire (SBQ). Where total daily sedentary behaviour ranges from 0 to 24 hours. Higher number of hours is worse.
Objectively measured total sedentary behaviour | Measured at week 0.
  Measured by the ACTIVPAL4
Objectively measured total sedentary behaviour | Measured at week 6.
  Measured by the ACTIVPAL4
Objectively measured total sedentary behaviour | Measured at week 12.
  Measured by the ACTIVPAL4

SECONDARY OUTCOMES:
Self-reported sedentary behaviour break frequency | Measured at week 0.
  Measured by the modified SIT-Q (no unabbreviated name) questionnaire. Where break frequency ranges from "less than every 30 minutes" to "over every 7 hours". Less frequent breaks is worse.
Self-reported sedentary behaviour break frequency | Measured at week 2.
  Measured by the modified SIT-Q (no unabbreviated name) questionnaire. Where break frequency ranges from "less than every 30 minutes" to "over every 7 hours". Less frequent breaks is worse.
Self-reported sedentary behaviour break frequency | Measured at week 4.
  Measured by the modified SIT-Q (no unabbreviated name) questionnaire. Where break frequency ranges from "less than every 30 minutes" to "over every 7 hours". Less frequent breaks is worse.
Self-reported sedentary behaviour break frequency | Measured at week 6.
  Measured by the modified SIT-Q (no unabbreviated name) questionnaire. Where break frequency ranges from "less than every 30 minutes" to "over every 7 hours". Less frequent breaks is worse.
Self-reported sedentary behaviour break frequency | Measured at week 12.
  Measured by the modified SIT-Q (no unabbreviated name) questionnaire. Where break frequency ranges from "less than every 30 minutes" to "over every 7 hours". Less frequent breaks is worse.
Self-reported sedentary behaviour break duration | Measured at week 0.
  Measured by the modified SIT-Q (no unabbreviated name) questionnaire. Where break duration ranges from "less than 30 seconds" to "over every 30 minutes". Shorter breaks are worse.
Self-reported sedentary behaviour break duration | Measured at week 2.
  Measured by the modified SIT-Q (no unabbreviated name) questionnaire. Where break duration ranges from "less than 30 seconds" to "over every 30 minutes". Shorter breaks are worse.
Self-reported sedentary behaviour break duration | Measured at week 4.
  Measured by the modified SIT-Q (no unabbreviated name) questionnaire. Where break duration ranges from "less than 30 seconds" to "over every 30 minutes". Shorter breaks are worse.
Self-reported sedentary behaviour break duration | Measured at week 6.
  Measured by the modified SIT-Q (no unabbreviated name) questionnaire. Where break duration ranges from "less than 30 seconds" to "over every 30 minutes". Shorter breaks are worse.
Self-reported sedentary behaviour break duration | Measured at week 12.
  Measured by the modified SIT-Q (no unabbreviated name) questionnaire. Where break duration ranges from "less than 30 seconds" to "over every 30 minutes". Shorter breaks are worse.
Self-reported screen time | Measured at week 0.
  Measured by a domain of the modified sedentary behaviour questionnaire (SBQ). Where total daily screen time ranges from 0 to 18 hours. Higher number of hours is worse.
Self-reported screen time | Measured at week 2.
  Measured by a domain of the modified sedentary behaviour questionnaire (SBQ). Where total daily screen time ranges from 0 to 18 hours. Higher number of hours is worse.
Self-reported screen time | Measured at week 4.
  Measured by a domain of the modified sedentary behaviour questionnaire (SBQ). Where total daily screen time ranges from 0 to 18 hours. Higher number of hours is worse.
Self-reported screen time | Measured at week 6.
  Measured by a domain of the modified sedentary behaviour questionnaire (SBQ). Where total daily screen time ranges from 0 to 18 hours. Higher number of hours is worse.
Self-reported screen time | Measured at week 12.
  Measured by a domain of the modified sedentary behaviour questionnaire (SBQ). Where total daily screen time ranges from 0 to 18 hours. Higher number of hours is worse.
Objective sedentary behaviour break frequency | Measured at week 0.
  Measured by the ACTIVPAL4
Objective sedentary behaviour break frequency | Measured at week 6.
  Measured by the ACTIVPAL4
Objective sedentary behaviour break frequency | Measured at week 12.
  Measured by the ACTIVPAL4
Objective sedentary behaviour break duration | Measured at week 0.
  Measured by the ACTIVPAL4
Objective sedentary behaviour break duration | Measured at week 6.
  Measured by the ACTIVPAL4
Objective sedentary behaviour break duration | Measured at week 12.
  Measured by the ACTIVPAL4
Self-reported quality of life | Measured at week 0.
  Measured by the modified short form -36 (SF-36) questionnaire. This questionnaire will use sub-scales: role limitations due to physical health (4 yes/ no questions), role limitations due to emotional problems (6 yes/no questions), energy, fatigue, and emotional well-being (9 six-point scale questions).
Self-reported quality of life | Measured at week 6.
  Measured by the modified short form -36 (SF-36) questionnaire. This questionnaire will use sub-scales: role limitations due to physical health (4 yes/ no questions), role limitations due to emotional problems (6 yes/no questions), energy, fatigue, and emotional well-being (9 six-point scale questions).
Self-reported quality of life | Measured at week 12.
  Measured by the modified short form -36 (SF-36) questionnaire. This questionnaire will use sub-scales: role limitations due to physical health (4 yes/ no questions), role limitations due to emotional problems (6 yes/no questions), energy, fatigue, and emotional well-being (9 six-point scale questions).
Overall experience of the intervention | Measured at week 6.
  The intervention group will receive at qualitative interview
Validate the modified sedentary behaviour questionnaire (SBQ) | Measured at week 0.
  The modified sedentary behaviour (SBQ) will be validated with the ACTIVPAL4
Validate the modified SIT-Q (no unabbreviated name) questionnaire | Measured at week 0.
  The modified SIT-Q (no unabbreviated name) questionnaires will be validated with the ACTIVPAL4
Validate the modified sedentary behaviour questionnaire (SBQ) | Measured at week 6.
  The modified sedentary behaviour (SBQ) will be validated with the ACTIVPAL4
Validate the modified SIT-Q (no unabbreviated name) questionnaire | Measured at week 6.
  The modified SIT-Q (no unabbreviated name) questionnaire will be validated with the ACTIVPAL4
Validate the modified sedentary behaviour questionnaire (SBQ) | Measured at week 12.
  The modified sedentary behaviour questionnaire (SBQ) will be validated with the ACTIVPAL4
Validate the modified SIT-Q (no unabbreviated name) questionnaire | Measured at week 12.
  The modified SIT-Q (no unabbreviated name) questionnaires will be validated with the ACTIVPAL4

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, PhD, Principal Investigator — Western University
Locations (1):
- Harry Prapavessis, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available to other researchers.